CLINICAL TRIAL: NCT04142463
Title: CONTACT-2: A Prospective Interventional Multicentre Before-after Study for the Implementation of a Care Pathway to Increase Self-management of Patients With Cancer Who Are Treated With Oral Anticancer Drugs
Brief Title: Collaborative Network to Take Responsibility for Oral Anticancer Therapy 2
Acronym: CONTACT-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ilyse Kenis (Other)
Collaborators: Kom Op Tegen Kanker (Other); KU Leuven (Other); University Ghent (Other)
Responsible Party: Sponsor-Investigator, Ilyse Kenis, PhD Researcher, KU Leuven
Organization: KU Leuven (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IK20082019
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Oncologic Disorders
Keywords: Oral anticancer drugs; Self-management; Care pathway; Before-after study; Self-management support
MeSH Terms: interventions — Critical Pathways

STUDY DESIGN:
Intervention Model Description: Patients will be recruited in phase 3 of the study, i.e. before the implementation of the care pathway (before-group) and in phase 6, i.e. after the implementation of the care pathway (after-group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before-group (No Intervention): This arm comprises patients who are recruited in phase 3 of the study, i.e. before the implementation of the care pathway. It is intended that patients included in phase 3 serve as a control-group for patients included in phase 6.
- After-group (Experimental): This arm comprises patients who are recruited in phase 6 of the study, i.e. after the implementation of the care pathway.
  Interventions: Other: Care pathway

INTERVENTIONS:
Other: Care pathway — A care pathway is a complex intervention for the mutual decision-making and organisation of care processes for a well-defined group of patients during a well-defined period. Care pathways can be used to optimise care processes when problems arise on communication, coordination, standardisation and monitoring of care for a specific group of patients. A care pathway for patients treated with OACD, should therefore consist of all relevant sustainable interventions that cover the continuum of the medicines' pathway with the aim to support self-management (e.g. consultations with doctors, contact moments with nurses, telephone follow-up, ...). The role of each stakeholder in the different interventions should be well-described including communication strategies between HCPs from primary and secondary care.
  Arms: After-group

SUMMARY:
In 2015, the research team of KU Leuven and UGent started a pilot project supported by Kom op Tegen Kanker, called CONTACT-1. This multicentre before-after study aims at developing, implementing and evaluating a care pathway for patients treated with oral anticancer drugs (OACD) in four oncology centres in Flanders (AZ Groeninge Kortrijk, AZ Imelda Bonheiden, AZ Maria Middelares Gent, AZ Turnhout).

Preliminary results from CONTACT-1 have shown that re-organisation of care processes, and better interdisciplinary collaboration and communication, are highly needed, and that working towards a care pathway is an appropriate method to achieve this. However, the development and implementation of the care pathway in each hospital was difficult and needed intensive coaching by the research team. Moreover, we have currently no insight in the impact of the care pathway on defined outcomes, neither on the sustainability of the implemented care pathway.

In CONTACT-2, we will expand the development and implementation of a care pathway to 10 additional oncology centres in Flanders. In contrast to CONTACT-1, the CONTACT-2 oncology centres will take the lead in the development, implementation and evaluation of the care pathway, supported by the research team en by the CONTACT-Toolkit. This toolkit was developed based on the experiences from CONTACT-1 and international guidelines on the implementation of care pathways/complex interventions.

Similar to CONTACT-1, we hypothesise that the implementation of a care pathway will improve the level of self-management and the quality of patient-centred care, and will increase adherence, patient satisfaction and health-related quality of life. Next, we hypothesise that the care pathway will improve counselling practice, interdisciplinary collaboration, self-efficacy and self-confidence of healthcare professionals (HCP). The impact of a care pathway on the above outcomes in patients as well as in HCPs will be investigated by means of various assessments, that have been selected by the research team based on their experiences from CONTACT-1. Moreover, we hypothesize that the development and implementation process will be more efficient in the CONTACT-2 oncology centres, who will need less intensive support of the research team, due to the CONTACT-Toolkit. A process evaluation will be conducted to test this last hypothesis.

Further in-depth analysis of the impact of the care pathway, combined with a thorough process evaluation, should eventually lead to insight in the crucial factors for sustainable implementation of a care pathway, as well as to definite conclusions on its impact for patients and HCPs.

Throughout CONTACT-2, the CONTACT-toolkit will be further elaborated, optimised and digitised based on the experiences of the research team and feedback from the CONTACT-2 oncology centres. The toolkit will enable a nation-wide and sustainable implementation of similar care pathways for patients treated with OACD.

DETAILED DESCRIPTION:
The study will be a prospective interventional multicentre before-after study with a total duration of 36 months and will be coordinated by a consortium of researchers from UGent and KU Leuven supported by Kom op Tegen Kanker. The intervention is the self-directed development and implementation of a care pathway in ten hospitals in Flanders.

The general lead throughout the study will be the 7-phase model for the development of a care pathway, which is translated to the specific context of OACD in the CONTACT-Toolkit. This methodology aims to offer a systematic approach for the support of an interdisciplinary team in the development of new care pathways or in the improvement of existing ones.

The CONTACT-Toolkit will serve as a roadmap that will guide the participating hospitals through the various phases and will therefore enable the self-directed development and implementation of the care pathway. Besides an overall guidance through the different phases of the 7-phase model, the toolkit contains additional tools including: presentations to structure internal meetings, tools and methods to map current practice, tools to measure key performance indicators, tools to support the development of a care pathway and tools to support counselling of patients treated with OACD (e.g. guide for telephone follow-up, guide for counselling at the start of the treatment).

In phase 1 and 2, a project structure is set up in each participating hospital by appointing a local coordinator and project team for the development of the care pathway. In phase 3, a detailed mapping of the current care process, which serves as before-study, will take place. Current practice will be evaluated from four different perspectives: own organisation and team, patients, external partners and independent observer. Assessments are performed by means of validated questionnaires and observations of daily practice by the research team. In phase 4, the care pathway will be developed by the project team, with respect to the results obtained from the mapping of current practice. During this phase, the research team will also provide training (i.e. e-learning, live training sessions) to all participating HCPs, to expand their medical knowledge on OACD and to improve counselling skills. The actual implementation of the care pathway is foreseen in phase 5. In phase 6, an evaluation of the care will be performed from the same four perspectives as in phase 3. This evaluation will include validated questionnaires, an interview with the coordinator, a focus group with the project team and participating HCPs and a second round of observations using a checklist and time task matrix of the care pathway document. In phase 7, the research team will take the necessary steps to guarantee the continuous follow-up of the care pathway without their further support.

To assess the impact of the care pathway on the level of the patient and the HCP, data obtained from the assessments in phase 3 (i.e. before-group) and 6 (i.e. after-group) will be compared. Furthermore, a process evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* A solid tumor and/or a haematological cancer
* Treated with one or more OACD (registered, "medical need" of "compassionate use")
* Able to swallow or retain oral medication

Exclusion Criteria:

* Following an adjuvant hormonal therapy with OACD (e.g. tamoxifen for 5 or 10 years)
* Following a therapy with a study drug in a phase I, II or III clinical trial
* Not able to understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in self-management | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  The ability of an individual to manage the symptoms, treatment, physical and psychosocial consequences and life style changes due to his/her condition. Adequate self-management refers to the ability to monitor one's condition and to effect cognitive, behavioural and emotional responses necessary to maintain a satisfactory quality of life.
  Questionnaire/method: Patient Activation Measure (PAM)

SECONDARY OUTCOMES:
Change in adherence | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  Questionnaire/method: Probabilistic Medication Adherence Scale (ProMAS)
Change in patients' experience with information on OACD | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  Questionnaire/method: Satisfaction with Information about Medicines Scale (SIMS)
Change in Health Related Quality of Life | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  Questionnaire/method: Functional Assessment of Cancer Therapy - General
Change in quality of patient-centred care | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  Questionnaire/method: CONTACT Patient-Centred Care Evaluation Questionnaire (PCCEQ)

OTHER OUTCOMES:
Change in clinician's beliefs on self-management | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  Questionnaire/method: Clinician Support for Patient Activation Measure (CS PAM)
Change in self-efficacy in HCPs | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  Questionnaire/method: Self-Efficacy and Performance in Self-management Support instrument (SEPSS-36)
Change in interdisciplinary collaboration | At baseline (before implementation of the care pathway); After 24 months (after implementation of the care pathway)
  Questionnaire/method: Clinician Staff Questionnaire (CSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Foulon, Prof. Dr., Principal Investigator — KU Leuven
Locations (10):
- Belgium (10):
  - AZ Klina Brasschaat, Brasschaat, Antwerpen
  - UZA, Edegem, Antwerpen
  - ZNA Jan Palfijn, Merksem, Antwerpen
  - H. Hartziekenhuis Mol, Mol, Antwerpen
  - Sint-Trudo ziekenhuis Sint-Truiden, Sint-Truiden, Limburg
  - AZ Vesalius Tongeren, Tongeren, Limburg
  - AZ Glorieux Ronse, Ronse, Oost-Vlaanderen
  - AZ Jan Portaels Vilvoorde, Vilvoorde, Vlaams-Brabant
  - AZ Sint-Lucas Brugge, Bruges, West-Vlaanderen
  - ZNA Middelheim, Antwerp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kinnaer LM, Decoene E, Van Hecke A, Foulon V. Collaborative network to take responsibility for oral anticancer therapy (CONTACT): Study-protocol investigating the impact of a care pathway. J Adv Nurs. 2019 Dec;75(12):3726-3739. doi: 10.1111/jan.14157. Epub 2019 Aug 27. PMID 31310353